CLINICAL TRIAL: NCT02252432
Title: Intraoperative Ketamine and Methadone for Laminectomy: Effect on Recovery, Postoperative Pain, and Opioid Requirements
Brief Title: The Effects of Ketamine and Methadone on Postoperative Pain for Laminectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No enough recruitments, very slow enrollment over the years
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00030109
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Laminectomy
Keywords: KETAMINE; METHADONE; POSTOPERATIVE PAIN; OPIOID REQUIREMENTS; Length of hospital stay; Perioperative outcomes
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine (Active Comparator): A bolus of intravenous (IV) ketamine during induction (0.5mg/kg), and an IV infusion of ketamine intraoperatively (5 mcg/kg/min))
  Interventions: Drug: Methadone; Drug: Ketamine + methadone
- Methadone (Active Comparator): Will receive a single dose of IV methadone (0.2 mg/kg) preinduction
  Interventions: Drug: Ketamine; Drug: Ketamine + methadone
- Ketamine + methadone (Experimental): Methadone (0.2 mg/kg) preinduction, a bolus of IV ketamine (0.5 mg/kg) during induction and IV ketamine infusion intraoperatively (5 mcg/kg/min)
  Interventions: Drug: Ketamine; Drug: Methadone

INTERVENTIONS:
Drug: Ketamine — A bolus of intravenous (IV) ketamine during induction (0.5mg/kg), and an IV infusion of ketamine intraoperatively (5 mcg/kg/min)
  Arms: Ketamine + methadone; Methadone
Drug: Methadone — A single dose of IV methadone (0.2 mg/kg) preinduction.
  Arms: Ketamine; Ketamine + methadone
Drug: Ketamine + methadone — Methadone (0.2 mg/kg) preinduction, a bolus of IV ketamine (0.5 mg/kg) during induction and IV ketamine infusion intraoperatively (5 mcg/kg/min)
  Arms: Ketamine; Methadone

SUMMARY:
The purpose of this research is to determine the pain-reducing effects of ketamine (Ketalar, an FDA-approved drug for anesthesia) and methadone (Dolophine, a long-acting narcotic) after lumbar laminectomy. The investigators would like to evaluate whether intraoperative use of both drugs may be able to provide better control of pain after lumbar surgery.

DETAILED DESCRIPTION:
During and after the surgery, patients undergoing surgery most likely need narcotics (opioids) that can cause side effects such as drowsiness and constipation. This can delay your recovery. The investigator would like to determine if the intraoperative use of ketamine and methadone will provide better pain control and reduce the use of narcotic painkiller medications (analgesics) after lumbar surgery as compared to either drug (ketamine or methadone) alone.

Ketamine is used to help to reduce the amount of the commonly used intravenous anesthetic drugs, minimize heart rate and blood pressure instability during surgery, and to improve outcomes after surgery (e.g. less pain, less constipation, less nausea and vomiting after surgery, faster return of bowel function and shortened length of hospital stay).

Ketamine is approved by the U.S. Food and Drug Administration (FDA) to be used: as an anesthetic and analgesic (painkiller). Ketamine is an "adjuvant," which is a drug that may increase the effectiveness or strength of other drugs when given at the same time. Ketamine is administered as an adjuvant during anesthesia to produce anesthetic and analgesic-sparing effects (reduce the amount of anesthetics and narcotics-painkiller drugs), hemodynamic stability (to maintain the blood pressure and heart rate within normal rank) and side effect reduction (e.g., constipation, nausea and vomiting, itching, and urinary retention). Ketamine will be used as approved in this study. Ketamine is frequently used intraoperatively for pain control in patients undergoing spine surgery at our institution and is within the standard of care. The standard of care indicates that this is one possible method which has been demonstrated to be safe and effective for patient care. This may vary at different institutions.

Methadone is approved by the U.S. Food and Drug Administration (FDA) to be used: as an opioid pain reliever, similar to morphine, and for narcotic detoxification to reduce withdrawal symptoms. The dose of methadone that will be used in this study may be slightly higher than the approved dose depending on the subject's weight. However, this dose of methadone is frequently used intraoperatively for pain control in patients undergoing spine surgery at our institution and is within the standard of care. This may vary at different institutions.

ELIGIBILITY:
Inclusion Criteria:

• 18 - 80 years old of either gender, scheduled for elective lumbar laminectomy

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) IV and above
* Intolerance, allergy, or contraindication to use of any medications used in this study
* Significant coronary artery disease (abnormal stress test, myocardial infarction

  * within the last 3 months)
* Increased intraocular pressure (e.g., untreated glaucoma)
* Uncontrolled hypertension (BP > 140/90)
* Sleep apnea and currently on continuous positive airway pressure (CPAP)
* Increased intracranial pressure or clinical signs thereof
* History of intracranial surgery, stroke, or brain aneurysm
* Cardiac arrhythmias particularly prolonged QT syndrome
* Drugs known to cause prolonged qT: class (IA) antiarrhythmics (quinidine, procainamide, disopyramide), class III antiarrhythmics (sotalol, dofetilide, ibutilide, amiodarone), haloperidol, thioridazine, arsenic trioxide, HIV protease inhibitors, tricyclic antidepressants
* Individuals with significant psychological disorders including: schizophrenia, mania, bipolar disorder or psychosis
* Pregnant or lactating women
* Emergent laminectomy
* Those already receiving ketamine or methadone prior to surgery
* Morbid obesity (BMI > 40 kg/m2) AND/OR weight > 150 kg
* Chronic renal failure ( creatinine > 2.0 mg/dL)
* Liver failure e.g., active cirrhosis
* Alcohol or substance abuse within in the past 3 months
* Uncorrected hypokalemia, hypomagnesemia, hypocalcemia (can be due to diuretics, mineralocorticoid use, laxatives)
* Chronic obstructive pulmonary disease (COPD)/Hypercarbia
* Restrictive lung disease (pulmonary fibrosis, myasthenia gravis)
* Congestive heart failure
* Thyroid disease
* Organ transplant patients
* Drugs/substances known to inhibit methadone metabolism: macrolide antibiotics e.g., erythromycin, cimetidine, astemizole, voriconazole, grapefruit juice

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, M.D., PhD., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
Started | 5 | 6 | 2
Completed | 5 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Methadone | Ketamine + Methadone | Total
Number analyzed (Participants) | 5 | 6 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 4 | 5 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 2 | 4 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 2 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption Obtained From the Recorded Data
Description: Perioperative use of opioid consumption inside the hospital (recorded by study staff and data obtained from patient charts)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
Number analyzed (Participants) | 5 | 6 | 2
milligram morphine equivalents | 23 (20) | 30 (16) | 26 (40)

2. Primary Outcome: Postoperative Pain
Description: Postoperative pain was measured at PACU using a Verbal Rating Scale from 0 to 10.
  Where 0= no pain and 10= maximum pain experienced
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
Number analyzed (Participants) | 5 | 6 | 2
score on a scale | 3.3 (2) | 4.1 (1) | 4.0 (1.2)

3. Secondary Outcome: Nausea and Vomiting
Description: The number of participants who experienced nausea and vomiting
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
Number analyzed (Participants) | 5 | 6 | 2
Participants | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Constipation at Follow up
Description: Day one, day three after surgery
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
Number analyzed (Participants) | 5 | 6 | 2
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: six weeks
Arm/Group | Ketamine | Methadone | Ketamine + Methadone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT02252432/Prot_SAP_000.pdf